CLINICAL TRIAL: NCT04924621
Title: Conventional Sedation Compaired With THRIVE Under General Anesthesia in Endotracheal Intubation by Fiberbronchoscope in Patients With Difficult Airways，A Randomized Controlled Study
Brief Title: Sedation Compaired With Anesthesia With THRIVE in Endotracheal Intubation With Difficult Airways
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, Chief of Department of Anesthesiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKUSSIRB-202163045
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Sedative, Hypnotic, or Anxiolytic Withdrawal; Airway Control
Keywords: Moderate Sedative; Airway Control; THRIVE
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE group (Experimental): Patients in group T received mask ventilation(oxygen concentration: 100%, flow rate: 6L /min, head height: 30°) for 5 minutes, and then THRIVE device (device model: Respiratory Humidification Treatment Device, AIRVO 2 PT101AZ, Fisher & Paykel Healthcare, Inc.) was set 100% oxygen, flow rate 30L /min, temperature 34℃.
  Interventions: Device: Respiratory Humidification Treatment Device, AIRVO 2 PT101AZ, Fisher & Paykel Healthcare, Inc.; Drug: Midazolam(T group); Drug: Sufentani(T group); Drug: Propofol(T group); Drug: Rocuronium(T group); Drug: Drug use target(T group)
- Control group (Placebo Comparator): The Control Group will receive mask ventilation (oxygen concentration: 100%, flow rate: 6L /min, head height: 30°) for 5 minutes
  Interventions: Device: Mask ventilation; Drug: Sufentanil(C group); Drug: Midazolam(C group); Drug: Propofol; Drug: Tetracaine(C group); Drug: Drug use target

INTERVENTIONS:
Device: Respiratory Humidification Treatment Device, AIRVO 2 PT101AZ, Fisher & Paykel Healthcare, Inc. — The nasal cavity was disinfected with Iodophor cotton swab, and the appropriate nasal cavity was selected for endotracheal intubation assisted by fiberoptic bronchoscope according to the experience of anesthesiologists.
  After the endotracheal intubation was fixed, the anesthesia machine was connected for mechanical ventilation. The anesthesia machine was set at 50% oxygen +50% air, and the tidal volume was set at 6-8ml/kg.
  Arms: THRIVE group
Device: Mask ventilation — The Control Group will receive sequential intravenous infusion of Sufentanil 5ug, midazolam 0.05mg/kg, and propofol 1-2ug/ml, to make the BIS between 70 and 80. 2ml tetracaine was injected with cyclothyroid membrane puncture, and the nasal cavity was disinfected with iodophor cotton swab. According to the experience of anesthesiologists, the appropriate nasal cavity was selected for intranasal endotracheal intubation assisted by fiberbronchoscope. After the endotracheal intubation was successful, the anesthesia machine was connected for mechanical ventilation, full narcotic inducer will be injected. The anesthesia machine was set at 50% oxygen +50% air, and the tidal volume was set at 6-8ml/kg.
  Arms: Control group
Drug: Midazolam(T group) — Midazolam 0.05mg/kg, intravenous injection
  Arms: THRIVE group
Drug: Sufentani(T group) — Sufentanil 0.02-0.05ug/kg, intravenous injection
  Arms: THRIVE group
Drug: Propofol(T group) — Propofol 2-3ug/ml, intravenous injection
  Arms: THRIVE group
Drug: Rocuronium(T group) — Rocuronium 0.06mg/kg, intravenous injection
  Arms: THRIVE group
Drug: Drug use target(T group) — Make BIS < 60 .
  Arms: THRIVE group
Drug: Sufentanil(C group) — Sufentanil 5ug, intravenous injection
  Arms: Control group
Drug: Midazolam(C group) — Midazolam 0.05mg/kg, intravenous injection
  Arms: Control group
Drug: Propofol — Propofol 1-2ug/ml, intravenous injection
  Arms: Control group
Drug: Tetracaine(C group) — 2ml tetracaine was injected with cyclothyroid membrane puncture.
  Arms: Control group
Drug: Drug use target — Make the BIS between 70 and 80.
  Arms: Control group

SUMMARY:
To compare the difference in endotracheal intubation in participants with difficult airway between under general anesthesia by Transnasal Humidified Rapid-Insufflation Ventilatory Exchange and under traditional sedation by mask ventilation. The investigators focus on the different outcomes in oxygenation maintaince, carbon dioxide removal and the effectiveness of safety apnea time, to evaluate the safety of receiving endotracheal intubation under general anesthesia in participants with difficult airway.

ELIGIBILITY:
Inclusion Criteria

* Age 18-60
* Patients with difficult airway assessed by two anesthesiologists according to the difficult airway score who needed to undergo nasal endotracheal intubation for oral and maxillofacial surgery in Peking University Stomatological Hospital.
* BMI between 18 to 30 kg/m2
* ASA Grade I to II
* NYHA grade I
* Patients requiring arterial hemodynamics monitoring and blood gas analysis due to surgical requirements
* Signed the informed consent

Exclusion Criteria

* Respiratory diseases: respiratory failure, COPD, pulmonary fibrosis, asthma and other diseases. Patients with ventilatory dysfunction or airway obstruction.
* NYHA cardiac function grade greater than I, or NYHA cardiac function grade I but with a history of coronary heart disease.
* Conditions affecting the monitoring of peripheral oxygen saturation, such as poor peripheral circulation perfusion and application of vasoconstrictor, are present.
* Indoor oxygen saturation below 92%.
* Patients who cannot tolerate rapid exchange ventilation with nasal humidification.
* Patients with a history of easy nasal bleeding.
* Inability to understand or express pain scores.
* Menstrual period and lactation period of female patients.
* The patient has mental illness.
* Patients with severe intraoperative complications should be removed after surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen pressure | Day 0
  Blood oxygen pressure after intubation immediately.
Pulse oxygen saturation | Day 0
  Pulse oxygen saturation after intubation immediately.
Blood carbon dioxide pressure | Day 0
  Blood carbon dioxide pressure after intubation immediately.

SECONDARY OUTCOMES:
Endtidal CO2 | Day 0
  Endtidal CO2 at time point of TA、TB、TC、TD
Success of intubation | Day 0
  Proportion of successful endotracheal intubation
Arrhythmias or dramatic haemodynamic fluctuations | Day 0
  Arrhythmias and dramatic fluctuations in heart rate and blood pressure: types and times of arrhythmias in the test were recorded. Changes in heart rate and blood pressure more than 30% before surgery were recorded as dramatic fluctuations.
Tolerance of intubation | Day 1
  The score of patient's tolerance to endotracheal intubation one day after surgery (0-10 points, 0 point is completely intolerable, 10 point is completely intolerable)
Time to complete intubation | Day 0
  Time required to complete endotracheal intubation
SPO2 below 95% | Day 0
  Percentage of patients with pulse oxygen saturation below 95% during the trial
SPO2 below 92% | Day 0
  Percentage of patients with pulse oxygen saturation below 92% during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No